CLINICAL TRIAL: NCT03758014
Title: A Randomized, Control, Open-label, Multicenter, Phase II/III Studies of Chlorogenic Acid for Injection for Safety and Efficacy of Grade IV GBM Patients
Brief Title: Studies of Chlorogenic Acid for Injection for Safety and Efficacy of Grade IV GBM Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan J.Z. Bio-chemical Science and Technology Development Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LYS-GBM-01
Record Dates: First submitted 2018-10-21; First posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: GBM
MeSH Terms: interventions — Chlorogenic Acid; Injections; Lomustine

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorogenic Acid for Injection (Experimental): 3 mg/kg per day, injection for 28 days，5 weeks per circle; max. 8 circles
  Interventions: Drug: Chlorogenic acid for Injection
- Lomustine (Active Comparator): 110 mg/m2 taken as a single oral dose every 6 weeks; max. 4 circles
  Interventions: Drug: Lomustine

INTERVENTIONS:
Drug: Chlorogenic acid for Injection — Chlorogenic acid (CHA) is a class 1 innovative small molecular natural drug, developed by Sichuan Jiuzhang Biological Science and Technology Co., Ltd. The mechanism of broad-spectrum antitumor activity is immunoregulation.
  Other Names: CHA
  Arms: Chlorogenic Acid for Injection
Drug: Lomustine — Lomustine (INN), abbreviated as CCNU (original brand name (formerly available) is CeeNU, now marketed as Gleostine), is an alkylating nitrosourea compound used in chemotherapy. It is closely related to semustine and is in the same family as streptozotocin. It is a highly lipid-soluble drug, thus it crosses the blood-brain barrier. This property makes it ideal for treating brain tumors, which is its primary use.
  Other Names: CCNU
  Arms: Lomustine

SUMMARY:
The purpose of phase II/III study: Determining the Overall Survival（OS）of Chlorogenic acid for injection comparing to in the advanced Glioblastoma Patients through study completion（an average of 18 months）after the first dose of chlorogenic acid for injection and Lomustine.

DETAILED DESCRIPTION:
Chlorogenic acid (CHA) is a class 1 innovative small molecular natural drug, developed by Sichuan Jiuzhang Biological Science and Technology Co., Ltd. The mechanism of broad-spectrum antitumor activity is immunoregulation. After received the clinical trial approval issued by CFDA, Jiuzhang Biotech successfully finished the phase I clinical studies of CHA for injection in advanced GBM patients, focus on safety, PK, and preliminary efficacy evaluation.

The results of phase I data showed that CHA had good safety, the main adverse effect was induration, no other serious adverse effects. PK exhibited that CHA had a rapid metabolism character (t1/2 = 1-1.5 h). In addition, there were no accumulative side effects for long-term use. To the investigators' surprise, the preliminary efficacy evaluation was amazing, there were 1 case CR and 1 case PR. The median OS of grade IV GBM patients was 21.4 months in effective dose group, which was much better than that of the historical reported data.The purpose of phase II/III study: Determining the Overall Survival（OS）of Chlorogenic acid for injection comparing to in the advanced Glioblastoma Patients through study completion（an average of 18 months）after the first dose of chlorogenic acid for injection and Lomustine .

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18;
2. KPS ≥ 60;
3. Recurrent GBM;
4. Estimated lifetime ≥ 3 months；
5. Female patients with negative pregnant test, and male/female patients of reproductive age without pregnancy planning in the next 12 months;
6. Volunteered for the phase 2 trial and sign the informed consent without protest.

Exclusion Criteria:

1. Patients who have received the therapy of chemotherapy or radical radiotherapy within 1 month before enrollment;
2. Pregnant or breast-feeding women, or patients(male and female) who have pregnancy plan;
3. Patients who had received a therapy of another investigational drug within 1 month；
4. Known active hepatitis B/hepatitis C, positive HIV/ syphilis antibody;
5. Patients who have received therapy of major surgery within 4 weeks or biopsy surgery within 1 week before enrollment;
6. Patient who need long term treatment of cortical hormone or other immunosuppressive drugs such as visceral organ transplanters；
7. Patients who have sufficient baseline organ function and whose laboratory data can meet the following criteria at the enrollment:1)PLT count<80×10~9/L； 2)NEUT# count<1.5×10~9/L ；3)HGB count<90g/L；4)Total bilirubin >1.5 times of ULN；5)ALT/AST >1.5 times of ULN；
8. History of drug abuse；
9. Patients who was treated with Immunologic drugs（DC/CIK/CTL/PD-（L）1） in 3 months;
10. Patients who are false progressers；
11. Patients who can not be received MRI examination；
12. Patients who had severe trauma or infectious diseases within 4 weeks；
13. Patients who had cerebral stroke or Transient ischemic attack within 6 months；
14. Patients who were performed important operations within 4 weeks；
15. Uncontrollable psychopaths;
16. Patients who had other advanced cancers within 5 years；
17. Patients who had grade III or IV heart failure within 6 months；
18. Other patients judged ineligible for enrollment in the study by the investigator (sub-investigator).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-11-27 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival（OS） | Through study completion（an average of 18 months）after the first dose of chlorogenic acid for injection and Lomustine

SECONDARY OUTCOMES:
progress free survival(PFS) | Through study completion（an average of 18 months）after the first dose of chlorogenic acid for injection and Lomustine
disease control rate（DCR) | Within the first 10 weeks after the first dose of chlorogenic acid for injection and Lomustine
objective response rate (ORR) | Within the first 10 weeks after the first dose of chlorogenic acid for injection and Lomustine
Karnofsky score standard | Through study completion（an average of 18 months）after the first dose of chlorogenic acid for injection and Lomustine
Montreal Cognitive Assessment score standard | Through study completion（an average of 18 months）after the first dose of chlorogenic acid for injection and Lomustine

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Li, Study Director — Beijing Tian Tan Hospital，Capital Medical University
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No